CLINICAL TRIAL: NCT02170116
Title: Pharmacodynamics, Safety and Pharmacokinetics After Single Oral Administration of 10, 30, 100, 200 and 400 mg BIBR 1048 MS as Drinking Solution in Healthy Subjects. An Open Study, Placebo Randomized Double Blind at Each Dose Level.
Brief Title: Pharmacodynamics, Safety and Pharmacokinetics After Oral Administration of BIBR 1048 MS in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1160.1
Record Dates: First submitted 2014-06-20; First posted 2014-06-23 (Estimated); Last update posted 2014-06-23 (Estimated); Status verified 2014-06

CONDITIONS: Healthy

ARMS (6):
- BIBR 1048 MS dose 1 (Experimental)
  Interventions: Drug: BIBR 1048 MS dose 1
- BIBR 1048 MS dose 2 (Experimental)
  Interventions: Drug: BIBR 1048 MS dose 2
- BIBR 1048 MS dose 3 (Experimental)
  Interventions: Drug: BIBR 1048 MS dose 3
- BIBR 1048 MS dose 4 (Experimental)
  Interventions: Drug: BIBR 1048 MS dose 4
- BIBR 1048 MS dose 5 (Experimental)
  Interventions: Drug: BIBR 1048 MS dose 5
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo to BIBR 1048 MS

INTERVENTIONS:
Drug: BIBR 1048 MS dose 1
  Arms: BIBR 1048 MS dose 1
Drug: BIBR 1048 MS dose 2
  Arms: BIBR 1048 MS dose 2
Drug: BIBR 1048 MS dose 3
  Arms: BIBR 1048 MS dose 3
Drug: BIBR 1048 MS dose 4
  Arms: BIBR 1048 MS dose 4
Drug: BIBR 1048 MS dose 5
  Arms: BIBR 1048 MS dose 5
Drug: Placebo to BIBR 1048 MS
  Arms: Placebo

SUMMARY:
The objective of this study was to assess safety, pharmacokinetics and the effect of BIBR 953 ZW on coagulation parameters of BIBR 953 ZW after oral single doses of the prodrug, BIBR 1048 MS, in healthy male subjects. This was the first administration of this substance to humans.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects as determined by results of screening
* Signed written informed consent in accordance with Good Clinical Practice (GCP) and local legislation
* Age >= 18 and <= 45 years
* Broca >= - 20 % and <= + 20 %

Exclusion Criteria:

* Any finding of the medical examination (including blood pressure, pulse rate and ECG) deviating from normal and of clinical relevance
* History or current gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunologic, hormonal disorders
* History of orthostatic hypotension, fainting spells or blackouts
* Diseases of the central nervous system (such as epilepsy) or psychiatric disorders
* Chronic or relevant acute infections
* History of

  * allergy/hypersensitivity (including drug allergy) which is deemed relevant to the trial as judged by the investigator
  * any bleeding disorder including prolonged or habitual bleeding
  * other hematologic disease
  * cerebral bleeding (e.g. after a car accident)
  * commotion cerebri
* Intake of drugs with a long half-life (> 24 hours) within 1 month prior to administration
* Use of any drugs which might influence the results of the trial within 10 days prior to administration or during the trial
* Participation in another trial with an investigational drug within 2 months prior to administration or during trial
* Smoker (> 10 cigarettes or 3 cigars or 3 pipes/day) or inability to refrain from smoking on study days
* Alcohol abuse (> 60 g/day)
* Drug abuse
* Blood donation within 1 month prior to administration or during the trial
* Excessive physical activities within 5 days prior to administration or during the trial
* Any laboratory value outside the clinically accepted reference range
* History of any familial bleeding disorder
* Thrombocytes < 150000/µl

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 1998-11; Primary Completion 1998-12 (Actual)

PRIMARY OUTCOMES:
Changes from baseline in prothrombin time (PT) (International Normalised Ratio (INR)) | - 0.5, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 hours after administration
Changes from baseline in activated partial thromboplastin time (aPTT) | - 0.5, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 hours after administration

SECONDARY OUTCOMES:
Peak (maximum) plasma concentration (Cmax) of BIBR 953 ZW | - 0.5, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48 hours after administration
time to reach the peak plasma concentration (tmax ) of BIBR 953 ZW | - 0.5, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48 hours after administration
AUC0-12 h - Area under the plasma concentration-time curve of BIBR 953 ZW from 0 to 12 h | - 0.5, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48 hours after administration
Area under the plasma concentration-time curve (AUC0-infinity) of BIBR 953 ZW from 0 to infinity | - 0.5, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48 hours after administration
Area under the plasma concentration-time curve of BIBR 953 ZW (AUCtf -infinity) from tf (last time point when measured plasma concentration) to infinity expressed as % of AUC0-infinity | - 0.5, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48 hours after administration
Terminal half-life(t1/2 ) of BIBR 953 ZW derived from non-compartmental analysis | - 0.5, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48 hours after administration
Total mean residence time (MRTtot ) of BIBR 953 ZW | - 0.5, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48 hours after administration
Total clearance (CLtot /f ) of BIBR 953 ZW after oral administration | 24 hours after administration
Volume of distribution (Vz/f ) of BIBR 953 ZW during terminal phase after oral administration | - 0.5, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48 hours after administration
Changes from baseline in Pulse rate | up to day 3
Changes from baseline in Systolic and diastolic blood pressure | up to day 3
Occurrence of Adverse events | up to day 3
Changes from baseline in Ecarin Clotting Time (ECT) | up to day 3
Changes from baseline in thrombin inhibition test time | up to day 3
Changes from baseline in thrombin time | up to day 3